CLINICAL TRIAL: NCT05864092
Title: Virtual Reality as an Adjuvant Therapy for Sickle Cell Vaso-Occlusive Crisis in the Pediatric Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UMMC-IRB-2023-8
Record Dates: First submitted 2023-04-24; First posted 2023-05-18 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Sickle Cell Crisis
Keywords: Virtual Reality; Sickle Cell Crisis
MeSH Terms: conditions — Vaso-Occlusive Crises

STUDY DESIGN:
Intervention Model Description: The study has two separate arms. A control arm will be a retrospective chart analysis of patients (100 anticipated) ages 6-21 with sickle cell VOC, and the trial arm will be an interventional prospective convenience sampling of patients (100 anticipated) admitted to the emergency department ages 6-21 with sickle cell VOC who will receive VR in addition to standard medical therapy.
Masking Description: Masking and randomization is not possible due to the nature of the virtual reality goggles.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): The control arm will be a retrospective chart review of patients ages 6 to 21 who present to the pediatric emergency department with sickle cell VOC listed as one of their diagnoses with the aim of identifying pain scores in accordance with medications received and identifying final disposition and identifying time in the emergency department and time to ED disposition. We aimed to review 100 charts. We found that 84 met inclusion criteria.
- Trial Arm (Experimental): The trial arm will be a prospective, convenience sampling of up to 100 patients ages 6 to 21 years who present to the pediatric emergency department with VOC listed as either their main complaint or as one of multiple complaints as identified by health care provider at time of presentation and meet inclusion criteria. The intervention will be virtual reality headset which will be offered simultaneously with standard medication therapy. We actually enrolled 17 patients who met inclusion criteria.
  Interventions: Other: Virtual Reality Goggles

INTERVENTIONS:
Other: Virtual Reality Goggles — We will offer patients virtual reality goggles with guided meditation software in addition to standard medical therapy (NSAID and opioid).
  Arms: Trial Arm

SUMMARY:
Vaso-occlusive crisis (VOC) is the most common complaint in patients with sickle cell disease presenting to the emergency room. VOC is most commonly treated with opioids and NSAIDs. However, new research is demonstrating that opioids in addition to virtual reality (VR) is more effective at reducing the experience of pain and pain nerve signals compared to opioids alone. Numerous research studies have demonstrated that VR reduces the experience of pain during painful medical procedures in children, such as venipuncture and burn wound dressing changes.

The study aims to add VR to standard of care medical treatment for pediatric patients with sickle cell disease who present to the pediatric emergency department in VOC. Investigators will conduct a retrospective chart review of patients aged 6 to 21 years with sickle cell disease who present to the pediatric emergency department with VOC for the historical control arm. Investigators will also conduct a prospective convenient sampling of patient who receive VR plus standard medical care in patients aged 6 to 21years with sickle cell disease who present to the emergency department with VOC. Investigators hypothesize that VR, in addition to standard medical care, will reduce the experience of pain and hospital admissions compared to the historical control group (standard medical treatment).

DETAILED DESCRIPTION:
Aim 1: To examine the effectiveness of VR plus standard medical therapy in reducing the experience of pain in patients 6 to 21 years with sickle cell VOC who present to the emergency department (ED), compared to historical standard medical care alone. Hypothesis 1: Patients who receive VR in addition to standard medical therapy will report lower pain severity when compared to historical control patients who received standard medical therapy alone.

Aim 2: To examine the effectiveness of VR plus standard medical therapy in reducing hospital admission rates for patients 6 to 21 years with sickle cell VOC who present to the ED, compared to historical standard medical therapy alone. Hypothesis 2: Patients who receive VR in addition to standard medical therapy will have a decreased rate of admission to the hospital compared to historical control patients who received standard medical therapy alone.

Secondary Aim 1: To examine the effectiveness of VR plus standard medical therapy in reducing length of stay in the ED Secondary Hypothesis 1: Patients who receive VR plus standard medical therapy will have shorter stays in the ED when compared to historical control patients who received standard medical therapy alone.

Secondary Aim 2: To examine the effectiveness of VR plus standard medical therapy in reducing time to ED disposition. Secondary Hypothesis 2: Patients who receive VR plus standard medical therapy will have shorter time to ED disposition when compared to historical control patients who received standard medical therapy alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 6 to 21 years
2. Sickle cell disease, any genotype
3. Diagnosis of VOC
4. Pain score of 4 or greater

Exclusion Criteria:

1. Non-VOC pain (from acute illness or injury)
2. Fever
3. Respiratory distress or acute chest syndrome or cough
4. Complaints of headache/dizziness/nausea during visit
5. History of epilepsy or seizures

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 101 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Pain Scores | Pain scores will be measured during patient stay in the ED. This is variable based on patient treatment course. For the trial arm, virtual reality therapy and time study team will interact with the patient is estimated to be 30 min.
  Patient pain scores will be recorded from time of patient presentation, after each dose of pain medication, at time of patient disposition. For the trial arm, pain scores will also be documented before and after the application of virtual reality goggles with guided meditation. Pain scores will be measured with the Wong-Baker Faces Scale generally for children 10 and under or depending on developmental and cognitive ability of the child or on a numeric scale from 0 to 10 with 0 correlating to "no pain" and 10 correlating to "severe pain."
Patient Disposition | Time frame is variable based on patient treatment course. For the trial arm, virtual reality therapy and time study team will interact with the patient is estimated to be 30 minutes.
  Patient disposition (admitted to hospital or discharged from emergency department) will be recorded.

SECONDARY OUTCOMES:
Length of Stay in the Emergency Department | Time frame is variable based on patient treatment course. For the trial arm, virtual reality therapy and time study team will interact with the patient is estimated to be 30 minutes.
  Time from patient arrival in the emergency department to patient leaving the emergency department (either through hospital admission or discharge)
Time to Emergency Department Disposition | Time frame is variable based on patient treatment course. For the trial arm, virtual reality therapy and time study team will interact with the patient is estimated to be 30 minutes.
  Time from patient arrival in the emergency department to disposition decision (hospital admission or discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Maready, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arane K, Behboudi A, Goldman RD. Virtual reality for pain and anxiety management in children. Can Fam Physician. 2017 Dec;63(12):932-934. PMID 29237632
- [Background] Hoffman HG, Chambers GT, Meyer WJ 3rd, Arceneaux LL, Russell WJ, Seibel EJ, Richards TL, Sharar SR, Patterson DR. Virtual reality as an adjunctive non-pharmacologic analgesic for acute burn pain during medical procedures. Ann Behav Med. 2011 Apr;41(2):183-91. doi: 10.1007/s12160-010-9248-7. PMID 21264690
- [Background] Hoffman HG, Richards TL, Van Oostrom T, Coda BA, Jensen MP, Blough DK, Sharar SR. The analgesic effects of opioids and immersive virtual reality distraction: evidence from subjective and functional brain imaging assessments. Anesth Analg. 2007 Dec;105(6):1776-83, table of contents. doi: 10.1213/01.ane.0000270205.45146.db. PMID 18042882
- [Background] Won AS, Bailey J, Bailenson J, Tataru C, Yoon IA, Golianu B. Immersive Virtual Reality for Pediatric Pain. Children (Basel). 2017 Jun 23;4(7):52. doi: 10.3390/children4070052. PMID 28644422
- [Background] Hoffman HG, Doctor JN, Patterson DR, Carrougher GJ, Furness TA 3rd. Virtual reality as an adjunctive pain control during burn wound care in adolescent patients. Pain. 2000 Mar;85(1-2):305-9. doi: 10.1016/s0304-3959(99)00275-4. PMID 10692634
- [Background] Chan E, Hovenden M, Ramage E, Ling N, Pham JH, Rahim A, Lam C, Liu L, Foster S, Sambell R, Jeyachanthiran K, Crock C, Stock A, Hopper SM, Cohen S, Davidson A, Plummer K, Mills E, Craig SS, Deng G, Leong P. Virtual Reality for Pediatric Needle Procedural Pain: Two Randomized Clinical Trials. J Pediatr. 2019 Jun;209:160-167.e4. doi: 10.1016/j.jpeds.2019.02.034. Epub 2019 Apr 29. PMID 31047650
- [Background] Walther-Larsen S, Petersen T, Friis SM, Aagaard G, Drivenes B, Opstrup P. Immersive Virtual Reality for Pediatric Procedural Pain: A Randomized Clinical Trial. Hosp Pediatr. 2019 Jul;9(7):501-507. doi: 10.1542/hpeds.2018-0249. Epub 2019 Jun 3. PMID 31160472
- [Background] Gold JI, SooHoo M, Laikin AM, Lane AS, Klein MJ. Effect of an Immersive Virtual Reality Intervention on Pain and Anxiety Associated With Peripheral Intravenous Catheter Placement in the Pediatric Setting: A Randomized Clinical Trial. JAMA Netw Open. 2021 Aug 2;4(8):e2122569. doi: 10.1001/jamanetworkopen.2021.22569. PMID 34432011
- [Background] Agrawal AK, Robertson S, Litwin L, Tringale E, Treadwell M, Hoppe C, Marsh A. Virtual reality as complementary pain therapy in hospitalized patients with sickle cell disease. Pediatr Blood Cancer. 2019 Feb;66(2):e27525. doi: 10.1002/pbc.27525. Epub 2018 Oct 26. PMID 30362236